CLINICAL TRIAL: NCT05578287
Title: Disitamab Vedotin Combined With Tislelizumab, Low-dose Capecitabine and Celecoxib as Salvage Therapy for HER2-positive Metastatic Colorectal Cancer: a Phase II Trial (DETECT)
Brief Title: RC48 Plus Tislelizumab, Low-dose Capecitabine and Celecoxib for HER2-positive Metastatic Colorectal Cancer
Acronym: DETECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-26
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer
Keywords: Salvage therapy; HER-2 positive; HER-2 ADC; PD-1 inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — disitamab vedotin; tislelizumab; Capecitabine; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-HER2 (Experimental): Disitamab Vedotin (2mg/kg, once every 2 weeks), Tislelizumab (2mg/kg, once every 2 weeks) combined with low-dose capecitabine 0.5g bid chemotherapy and the COX2 inhibitor celecoxib 200mg bid as salvage therapy
  Interventions: Drug: Anti-HER2 ADC

INTERVENTIONS:
Drug: Anti-HER2 ADC — Disitamab Vedotin (2mg/kg, q2w), Tislelizumab (2mg/kg, q2w) combined with low-dose capecitabine 0.5g bid chemotherapy and the COX2 inhibitor celecoxib 200mg bid
  Other Names: Disitamab Vedotin; Tislelizumab; Capecitabin; Celecoxib

SUMMARY:
As an established therapeutic target, HER2 is widely used in a variety of tumors, including breast cancer and gastric cancer, among which a variety of drugs, including trastuzumab, lapatinib and T-DM1, have been approved for the treatment of breast cancer and gastric cancer with HER2 amplification or overexpression. In colorectal cancer, HER2 as a target has also been focused in recent years.

ELIGIBILITY:
Inclusion Criteria:

1. A voluntarily signed and dated informed consent must be obtained from the subject in accordance with regulations and institutional guidelines before performing any protocol-related procedures other than routine care;
2. Aged 18-75;
3. Patients with pathologically or cytologically confirmed adenocarcinoma of the colon or rectum with evidence of locally advanced lesions or metastases that could not be resected;
4. ECOG performance status score is 0-1;
5. Detection of HER2-positive tumor tissue at any time before screening; HER2 positive was defined as the presence of HER2 3+ positive staining in more than 50% of tumor cells on IHC. Or patients with a HER2 score of 2+ should also be tested by FISH: HER2/CEP17 ratio ≥2.0.
6. Appropriate organ function based on the following laboratory test values obtained during the screening period:

   Neutrophil count ≥1.5×109/L, platelet count ≥75×109/L, serum total bilirubin ≤ 1.5× upper normal limits, UNL), aspartate aminotransferase ≤ 2.5×UNL, alanine aminotransferase ≤ 2.5×UNL, serum creatinine ≤ 1.5×UNL;
7. Previous chemotherapy including oxaliplatin, irinotecan, and fluorouracil failed, including the following:

   Subjects using oxaliplatin as adjuvant therapy should have treatment progression within 6 months of completion of adjuvant therapy; Patients who refused standard chemotherapy because of unacceptable toxicity to treatment will be admitted to the study;
8. Previous or no previous anti-HER2-targeted therapy, disease progression or intolerable toxicity during or within 3 months after treatment;
9. Measurable lesions, according to the Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1;

Exclusion Criteria:

1. Complicated with intestinal obstruction, active bleeding or perforation and requiring emergency surgery;
2. Major surgery or severe trauma, such as laparotomy, thoracotomy, laparoscopic organ resection, etc. within the previous 4 weeks (the surgical incision should be completely healed before enrollment);
3. Had active coronary artery disease, severe/unstable angina pectoris or newly diagnosed angina pectoris or myocardial infarction in the 12 months prior to study enrollment;
4. Thrombotic or embolic events occurred within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, deep vein thrombosis;
5. The New York Heart Association (NYHA) class II or higher congestive Heart failure;
6. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; Hepatitis C, defined as HCV-RNA above the detection limit of the assay) or co-infection with hepatitis B and C;
7. The presence of any active, known or suspected autoimmune disease. To allow enrollment of subjects in stable condition who do not require systemic immunosuppressive therapy, such as type I diabetes, hypothyroidism that requires only hormone replacement therapy, and skin conditions that do not require systemic treatment (e.g., vitiligo, psoriasis, and alopecia);
8. The presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes mellitus, hypertension, pulmonary fibrosis, and acute pneumonia);
9. Common Terminology Criteria for Adverse events that have not resolved due to any previous treatment CTCAE) (version 5.0) grade 2 or higher toxicity (except peripheral neurotoxicity, anemia, alopecia, skin pigmentation);
10. Previous recipients of PD-1/PD-L1 inhibitors or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibodies;
11. A history of known or suspected allergies to any of the relevant drugs used in the study;
12. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Safety | 1 year
  Safety was assessed by evaluation of AEs and serious AEs according to CTCAE 5.0
Feasibility | 1 year
  Feasibility was determined based on any treatment -related AEs leading to delays over 15 days or discontinous of treatment.

SECONDARY OUTCOMES:
Objective response rate | 1 year
  The percentage of subjects with Complete Response (CR) and Partial Response (PR).
disease control rate,DCR | 1 year
  The percentage of subjects with total number of Complete Response (CR), Partial Response (PR) and stable disease (SD).
Progression-free survival (PFS) | 1 year
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first.
Overall Survival (OS) | 2 year
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided